CLINICAL TRIAL: NCT02993484
Title: The Role of Mitochondrial Respiration in the Cardioprotective Capacity of IPC in Diabetic and Non-diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Human A-strips Mitochondria
Record Dates: First submitted 2016-12-08; First posted 2016-12-15 (Estimated); Last update posted 2019-06-07 (Actual); Status verified 2018-10

CONDITIONS: Reperfusion Injuries, Myocardial
MeSH Terms: conditions — Myocardial Reperfusion Injury | interventions — methyl malonate; Ischemic Preconditioning; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- non-diabetic Sham control (Experimental): Heart tissue obtained from non-diabetic patients undergoing surgery will not receive drugs or ischemia
  Interventions: Other: Sham
- non-diabetic Ischemia reperfusion (Experimental): Heart tissue from non-diabetic patients undergoing surgery will not receive drugs but will receive ischemia
  Interventions: Other: Ischemia reperfusion
- non-diabetic Ischemic preconditioning (Experimental): Heart tissue from non-diabetic patients undergoing surgery will not receive drugs but will receive short periods of ischemia prior to index ischemia
  Interventions: Biological: Ischemic preconditioning
- non-diabetic Dimethyl malonate (Experimental): Heart tissue from non-diabetic patients undergoing surgery will receive a drug (Dimethyl Malonate) prior to index ischemia
  Interventions: Drug: Dimethyl Malonate
- Diabetic Sham control (Experimental): Heart tissue obtained from diabetic patients undergoing surgery will not receive drugs or ischemia
  Interventions: Other: Sham
- Diabetic Ischemia reperfusion (Experimental): Heart tissue from diabetic patients undergoing surgery will not receive drugs but will receive ischemia
  Interventions: Other: Ischemia reperfusion
- Diabetic Ischemic preconditioning (Experimental): Heart tissue from diabetic patients undergoing surgery will not receive drugs but will receive short periods of ischemia prior to index ischemia
  Interventions: Biological: Ischemic preconditioning
- Diabetic Dimethyl malonate (Experimental): Heart tissue from diabetic patients undergoing surgery will receive a drug (Dimethyl Malonate) prior to index ischemia
  Interventions: Drug: Dimethyl Malonate

INTERVENTIONS:
Drug: Dimethyl Malonate — Heart tissue will be obtained from patients undergoing heart surgery. The tissue will be used to test the properties of ischemia and different cardioprotective interventions.
  Other Names: Dimethyl Malonate; PubChem Substance ID 24848281
  Arms: Diabetic Dimethyl malonate; non-diabetic Dimethyl malonate
Biological: Ischemic preconditioning — Heart tissue will be obtained from patients undergoing heart surgery. The tissue will be used to test the properties of ischemia and different cardioprotective interventions.
  Arms: Diabetic Ischemic preconditioning; non-diabetic Ischemic preconditioning
Other: Ischemia reperfusion — Heart tissue will be obtained from patients undergoing heart surgery. The tissue will be used to test the properties of ischemia and different cardioprotective interventions.
  Arms: Diabetic Ischemia reperfusion; non-diabetic Ischemia reperfusion
Other: Sham — Heart tissue will be obtained from patients undergoing heart surgery. The tissue will be used to test the properties of ischemia and different cardioprotective interventions.
  Arms: Diabetic Sham control; non-diabetic Sham control

SUMMARY:
The overall aim of this study is to examine the role of mitochondrial respiration in human diabetic tissue before and after ischemia. Furthermore we will examine the ability of ischemic preconditioning (IPC) to preserve the mitochondrial function and hemodynamic performance of both non-diabetic and diabetic fibers after ischemia. To increase our understanding on the metabolic changes during ischemia in both non-diabetic and diabetic tissue we will use Dimethyl Malonate and examine the impact of this blockade on post-ischemic mitochondrial respiration.

DETAILED DESCRIPTION:
20 diabetic and 20 non-diabetic patients undergoing elective CABG surgery or other heart surgery where extracorporal circulation is used will be included in the study. The patiens will not be given any treatment prior to the operation. During the cardiac surgery a small sample of the heart is routinely removed when the patient is connection to the heart-lung machine. From this tissue sample it is possible to isolate muscle trabeculae which will be used in an atrial strip model and randomized to one of four types of treatment. Simultaneously with the isolation of the trabeculae, a fifth trabecular will be used to assess mitochondrial respiration at baseline. Group 1 will serve as a sham control, group 2 will serve as ischemic control and receive an extended period of hypoxia, Group 3 will be treated with ischemic preconditioning, where short periods of non lethal lack of oxygen will be given directly to the tissue (after removal from the patient) prior to the extended period of hypoxia, Group 4 will receive dimethyl malonate prior to the prolonged hypoxia.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing CABG or other surgery where extracorporal circulation will be used.

Exclusion Criteria:

* raise in ischemic markers within 4 weeks
* ejection fraction <30
* Atrial fibrilation
* Oral opioid treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-12; Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Mitochondrial respiration of individual complexes | Outcome will be assessed within a year when the inclusion of patients is complete
  Mitochondrial respiration of individual complexes will serve as primary outcome and will be examined by oxygraph technique.

SECONDARY OUTCOMES:
Hemodynamic performance | Outcome will be assessed within a year when the inclusion of patients is complete
  Hemodynamic performance will be measured as contractile force of heart fibers before during and after ischemia.

IPD SHARING:
Plan to Share IPD: No